CLINICAL TRIAL: NCT04919421
Title: Comparative Evaluation of The Analgesic Effect of Virtual Reality With Topical Anesthesia to Reduce Pain During Administration of Local Anesthesia
Brief Title: Comparison Between the Analgesic Effectiveness of Virtual Reality and Topical Anesthesia: A Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riyadh Elm University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RiyadhEU
Record Dates: First submitted 2019-10-30; First posted 2021-06-09 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Pain
Keywords: pain perception; virtual reality
MeSH Terms: conditions — Pain | interventions — Dental Health Services

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Virtual reality (Active Comparator): Participants will wear a virtual reality headset during the dental injection in which a video is playing.
  Interventions: Device: Dental injection and virtual reality device
- Topical gel (Active Comparator): Participants will receive application of topical anesthetic gel on the site of dental injection.
  Interventions: Drug: Dental injection and topical gel application

INTERVENTIONS:
Drug: Dental injection and topical gel application — Topical anesthesia gel will be applied followed by dental injection with 1.8 ml Xylocaine 20mg/ml (DENSPLY Pharmaceutical); adrenaline: 1 : 100.000, delivered in cartridges using a 27 -gauge short needle (0.4 x 25 mm,C-K jet) and sterile non-aspirating syringe.
  Other Names: No other name
  Arms: Topical gel
Device: Dental injection and virtual reality device — Dental injection will be made while the participants are wearing virtual reality device.
  Other Names: No other name
  Arms: Virtual reality

SUMMARY:
A split-mouth, controlled trial aimed to clinically compare and evaluate the effectiveness of virtual reality versus topical anesthesia gel prior to administration of dental anesthesia injection in reducing the perceived pain and anxiety level in adult patients and to find out their preferred procedure.

Heart rate before and after the end of the procedure will be identified, pain intensity of the injection will be identified using a scale, and finally patients' preference will be identified using a questionnaire.

DETAILED DESCRIPTION:
Steps of the Experiment

Step I: before the administration of the local anesthesia injection, heart rate will be measured for the patients using an FDA Approved pulse oximeter (Santa Medical SM-165 Finger Pulse Oximeter). Findings will be recorded.

Step II: at the first appointment, patients will be randomly allocated to receive the injection of the local anesthesia either with topical anesthetic gel or with virtual reality in one side of the jaw.

Step III: immediately after dental anesthesia injection procedure, the patient will be asked to rate the level of perceived pain, using Wong-Baker faces pain rating scale (WBFPS).

Step IV: after the administration of the local anesthesia injection, heart rate will be measured for the patients an FDA Approved pulse oximeter (Santa Medical SM-165 Finger Pulse Oximeter). Findings will be recorded.

Step V: in the next appointment, the other technique (virtual reality or topical anesthetic gel) will be used on the contralateral side for the same patients.

So each patient will receive local anesthesia injection twice, one with topical anesthetic gel and one else with VR in the contralateral side.

Step VI: after completion of both procedures, each patient will be asked to state his/her preference for the delivery system of future injections to be recorded.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) class I, aged between 18 and 65, both male and female, who required bilateral local anesthetic injections in the premolar teeth in the upper jaw.
* Participants are in good general health, take no medications, and have no contraindications to the use of local anesthetic.
* The ability to understand oral and written instructions, and the ability to use the VR controller.

Exclusion Criteria:

* Patients who need intravenous sedation cannot participate in the study.
* If a patient requires only single visit/ treatment or if he/she cannot attend the other visit.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-11-10 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Heart rate | immediately after the intervention/procedure (injection)
  heart rate will be measured for the participants using an FDA Approved pulse oximeter (Santa Medical SM-165 Finger Pulse Oximeter)
Wong-Baker faces pain rating scale (WBFPS) | 3 minutes after the intervention/procedure (injection)
  A tool to measure the intensity of pain comprising a scale from 0 to 10. The patient will select a number based on the intensity of the pain, "0" means no pain, "10" means extremely severe pain.
Participant's future preference | 5 minutes after the intervention/procedure (injection)
  Each participant will be asked by a questionnaire to state his/her preference for the delivery system of future injections

CONTACTS AND LOCATIONS:
Overall Officials: Ammar AbuMostafa, BDS, MSC, Study Director — Riyadh Elm University
Locations (1):
- Riyadh Elm University, Riyadh, Saudi Arabia

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-04-28): https://cdn.clinicaltrials.gov/large-docs/21/NCT04919421/Prot_SAP_ICF_000.pdf